CLINICAL TRIAL: NCT01601587
Title: Introduction Seminar About Patient Participation, Treatment Options and Decisional Preferences for Psychiatric Outpatients on Waiting List
Brief Title: Introduction Seminar About Patient Participation and Treatment Options Decisional Preferences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4.2009.77.2009/1980 ( part 2)
Record Dates: First submitted 2012-05-10; First posted 2012-05-18 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Mental Health Disorders
Keywords: Introductory Seminar; Waiting list; Community Mental Health Centre

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (No Intervention): Patients will receive treatment as usual
- Introduction Seminar (Other): Psychoeducational group
  Interventions: Other: A psychoeducational group intervention.

INTERVENTIONS:
Other: A psychoeducational group intervention. — The intervention is an introduction seminar. It will be held over FOUR hours. Up to 15 patients can participate in each seminar. The content of the was developed based on study 1. The presentation about available treatment options and patient's rights are made by multi professional health personnel and user representatives. More specifically, this will be done under the following topics:
  1. What is mental health?
  2. Treatment options: orientation about individual and group based treatment modalities.
  3. Former patients experience with their own treatment, self-help and participation.
  4. How to influence and participate actively in the treatment and patient rights.
  5. What can I do while I wait for treatment and where can I otherwise do to avoid aggravation?
  Arms: Introduction Seminar

SUMMARY:
Patient participation (PP) in Hospital is a goal defined by the Norwegian Health Authorities and it is a mandatory activity for District Psychiatric out-patient Centres (DPC) in Norway: patients are entitled to have influence on their treatment and should receive sufficient information directed at empowerment. Nevertheless, studies from Norway have found that patients who seek help are dissatisfied with the information they receive and doubt their possibility for real influence on their treatment. One way to improve individual PP might be to give patients sufficient information and education before they start their treatment in the form of an educational group intervention, an introduction seminar (IS); this group intervention is less time and resource consuming than individual interventions.

Aims: The main purpose of this project is to develop and evaluate an IS for patients on a waiting list of DPC. The seminar will educate patients, so they can actively participate in their own treatment and, thereby, choosing treatment, reducing the risk of dropping out of treatment. Another aim is to enable patients to participate in their own treatment, to cope with their problems while they are waiting for treatment by providing them contact with primary health care and user organizations during their waiting time, and to increase adherence.

Methods: The project involves three components: an exploratory study of educational content of the seminar; RCT of that 4-hours program (to examine its effect on treatment preferences and choices, activation, satisfaction, mental health and cost-benefit) and then a post-seminar qualitative evaluation, which will be used to create a broad yet deep understanding of the practical side of the participants'experience and the seminar's effect.

DETAILED DESCRIPTION:
Part I: An exploratory study of educational content of the seminar: a qualitative study (started october 2011)

Part II (RCT)

The intervention:

The introduction seminar will be held over one half day, 4 hours. Up to 15 patients can participate in each seminar. The content was developed based on study 1. The presentation about available treatment options and patient's rights are made by multi professional health personnel and user representatives. More specifically, this will be done under the following topics:

1. What is mental health?
2. Treatment options: orientation about individual and group based treatment modalities.
3. Former patients experience with their own treatment, self-help and participation.
4. How to influence and participate actively in the treatment and patient rights.
5. What can I do while I wait for treatment and where can I otherwise do to avoid aggravation?.

At the end of the day, the patients will be divided into small groups mentored by health personnel where they can discuss the presentations and ask questions. In the breaks, literature and other kinds of information for patients will be on display. All participants will get a folder with details of the program and leaflets from patient organisations and governmental agencies.

Sample size Selected Treatment: The number of patients is calculated based on a significance level of 5% and a power of 93%. The numbers needed in each group becomes 25 (calculated using IR), and the aim is to include a total of 52 patients in the RCT. It is controlled that it is feasible to recruit this number of patients.

PAM: Number of patients is calculated based on a significance level of 5% and a power of 87%. The standard deviation is estimated to be 13.8 and 9.7 (Pilot RCT data). The numbers needed in each group becomes 25 (calculated using SamplePower v2.0, SPSS Inc), and the aim is to include a total of 52 patients. It is controlled that it is feasible to recruit this number of patients.

Part III Qualitative and quantitative analysis:

To obtain information about the patients experience after the intervention, a post-seminar qualitative evaluation will be conducted:

15 randomly selected patients will additionally participate in the seminar, and they will be take part in Part III and in the quantitative part of the study.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* referred for out-patient treatment
* guarantee of starting treatment between 2 and 4 months

Exclusion Criteria:

* guarantee of starting treatment in less than 2 months
* Patients who do not understand the consequences of taking part of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Selected Treatment | 1 month
  one single question
Health Care utilization | 1 year
  Health care registration (adherence, attendance, consultations, dropout's rates and cost)
Health Care utilization | 2 years
  Health care registration (adherence, attendance, consultations, dropout's rates and cost)
coping | 4 months
  Patient Activation Measure (PAM-13)

SECONDARY OUTCOMES:
Preferences for involvement in treatment decision making | Baseline, 1, 4 and 12 months
  Control Preferences Scale
Treatment Satisfaction | Baseline, 1, 4, and 12 months
  Client Satisfaction Questionnaire-8 (CSQ-8)
Quality of Life | Baseline, 1, 4 and 12 months
  WHO-Five Well-being Index (WHO-5)
Motivation | Baseline, 1, 4 and 12 months
  One single question about motivation for treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Olav Linaker, md phd, Principal Investigator — National Taiwan Normal University
Locations (1):
- Tiller DPS, Trondheim, Norway

REFERENCES:
- [Result] Lara-Cabrera ML, Salvesen O, Nesset MB, De las Cuevas C, Iversen VC, Grawe RW. The effect of a brief educational programme added to mental health treatment to improve patient activation: A randomized controlled trial in community mental health centres. Patient Educ Couns. 2016 May;99(5):760-8. doi: 10.1016/j.pec.2015.11.028. Epub 2015 Dec 2. PMID 26682971